CLINICAL TRIAL: NCT02210429
Title: Supraclavicular Blocks for Post-Operative Pain Control in Supracondylar Fracture Fixation, a Retrospective Analysis of Single Shot Catheter Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2014-15849
Record Dates: First submitted 2014-08-03; First posted 2014-08-06 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-06

CONDITIONS: Acute Pain; Pain, Postoperative
Keywords: Supraclavicular Block; Supraclavicular Catheter; Pediatric Anesthesia; Regional Anesthesia; Supracondylar Elbow Fracture
MeSH Terms: conditions — Acute Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IV Opioids (Active Comparator)
  Interventions: Procedure: Elbow Fracture Fixation
- Supraclavicular Single-Shot Block (Active Comparator)
  Interventions: Procedure: Elbow Fracture Fixation
- Supraclavicular Catheter (Active Comparator)
  Interventions: Procedure: Elbow Fracture Fixation
- Supraclavicular Angiocath (Active Comparator)
  Interventions: Procedure: Elbow Fracture Fixation

INTERVENTIONS:
Procedure: Elbow Fracture Fixation

SUMMARY:
We hypothesize that patients who receive a supraclavicular block via Angiocath, placed intra-operatively and dosed post-operatively following neurologic examination, will have lower pain scores, lower use of intravenous morphine equivalents in the post-anesthesia care unit, and lower rates of intervention for post-operative nausea and vomiting. We also hypothesize that patients receiving this nerve block had the same rates of nerve damage as the patients who did not receive a block and that there will be no demonstrable safety concerns with this block.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18
* Undergoing supracondylar fracture fixation in operating room

Exclusion Criteria:

* Incomplete or inaccessable chart data

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative opioid use | 24 hours
  Total doses

SECONDARY OUTCOMES:
Anti-emetic drug use | 24 hours
  Total doses
Incidence of nerve damage or compartment syndrome | 1 month
  Evaluated by surgeon at follow up.
Pain Score | 24 hours
  Using Visual Analog Scale and FLACC pain scale (for younger children) we will compare pain scores in the various groups.

CONTACTS AND LOCATIONS:
Overall Officials: Santhanam Suresh, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Suresh S, Sarwark JP, Bhalla T, Janicki J. Performing US-guided nerve blocks in the postanesthesia care unit (PACU) for upper extremity fractures: is this feasible in children? Paediatr Anaesth. 2009 Dec;19(12):1238-40. doi: 10.1111/j.1460-9592.2009.03182.x. No abstract available. PMID 20017868
- [Background] Steinfeldt J, Robison T, Przybylo HJ. Placement of an US-guided supraclavicular block postoperatively in children: can we make this easy? Paediatr Anaesth. 2010 Aug;20(8):780-1. doi: 10.1111/j.1460-9592.2010.03355.x. No abstract available. PMID 20670249